CLINICAL TRIAL: NCT00392444
Title: A Phase II Study of Sunitinib (SU11248; NSC 736511; IND 74019) in Patients With Advanced Malignant Pleural Mesothelioma
Brief Title: Sunitinib in Treating Patients With Advanced Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00693; NCI-2009-00693 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000652058; NCIC-183 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-183 (Other: CTEP)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Malignant Mesothelioma; Recurrent Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with advanced malignant mesothelioma of the pleura. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of sunitinib malate, in terms of response rate (complete and partial), in patients with malignant pleural mesothelioma.

II. Assess the toxicity, safety, and tolerability of this drug in these patients.

III. Assess the duration of response or stable disease, stable disease rate, progression-free survival, and median and overall survival rates.

OUTLINE: This is a multicenter, nonrandomized, open-label study. Patients are stratified according to prior cytotoxic chemotherapy (yes vs no).

Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Criteria:

* Histologically or cytologically confirmed malignant pleural mesothelioma; Advanced or metastatic disease incurable by standard therapies
* Measurable disease, defined as at least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan; No sole site of disease in a previously irradiated area unless there has been subsequent evidence of progression; Low-dose, palliative radiotherapy allowed
* Meets 1 of the following criteria for prior cytotoxic chemotherapy treatment: Previously treated with 1 platinum-based chemotherapy regimen; Previously untreated (i.e., no prior cytotoxic chemotherapy)
* No known brain metastases
* ECOG performance status 0-1
* Life expectancy >= 12 weeks
* Platelet count >= 100,000/mm^3
* Absolute granulocyte count >= 1,500/mm^3
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Calcium =< 3 mmol/L
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients must reside within a 1.5 hour drive from participating center
* Able to take oral medication
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer, curatively treated in-situ carcinoma of the cervix, or any other curatively treated solid tumor
* No known history of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* No QTc prolongation (i.e., QTc interval >= 500 msec) or other significant ECG abnormalities
* No New York Heart Association (NYHA) class III or IV heart failure
* Patients with the following histories allowed provided they are asymptomatic with respect to cardiac function and LVEF is normal by MUGA at baseline: Anthracycline exposure, Central thoracic radiation that included the heart, NYHA class II cardiac function
* No uncontrolled hypertension (i.e., systolic blood pressure >= 140 mm Hg or diastolic blood pressure >= 90 mm Hg)
* No cardiac disease within the past 12 months, including any of the following: myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure
* No pulmonary embolism within the past 12 months
* No cerebrovascular accident or transient ischemic attack within the past 12 months
* No bowel obstruction or any condition that would impair the ability to swallow and retain sunitinib malate, including any of the following:

gastrointestinal tract disease resulting in an inability to take oral medication, requirement for IV alimentation, active peptic ulcer disease

* No serious illness or medical condition that would preclude study treatment including, but not limited to, any of the following: history of significant neurologic or psychiatric disorder that would impair the ability to obtain consent or limit compliance with study requirements, Active uncontrolled infection, Any other medical condition that might be aggravated by treatment, OR;
* Serious or nonhealing wound, ulcer, or bone fracture, Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No pre-existing hypothyroidism unless euthyroid on medication
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following: Azole antifungals (e.g., ketoconazole, itraconazole, miconazole), Verapamil, Clarithromycin, HIV protease inhibitors (e.g., indinavir, saquinavir, ritonavir, atazanavir, or nelfinavir) Erythromycin, Delavirdine, Diltiazem
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following: Rifampin, Phenytoin, Rifabutin, Hypericum perforatum (St. John's wort), Carbamazepine, Efavirenz Phenobarbital, Tipranavir
* At least 4 weeks since prior major surgery and recovered
* At least 4 weeks since prior radiotherapy and recovered
* At least 12 months since prior coronary/peripheral artery bypass graft or stenting
* No prior surgical procedures affecting absorption
* No prior radiotherapy that involved >= 30% of functioning bone marrow
* No prior treatment with any other antiangiogenic agents or multitargeted tyrosine kinase inhibitors, including any of the following:

bevacizumab, sorafenib tosylate, pazopanib, thalidomide, AZD2171, vandetanib, AMG706, vatalanib, VEGF Trap

* No prior angiogenesis inhibitors except epidermal growth factor receptor inhibitors or other noncytotoxic therapy
* No other concurrent anticancer therapy or treatment with other investigational anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic doses of coumadin-derivative anticoagulants (e.g., warfarin); Doses =< 2 mg/day for prophylaxis of thrombosis or low molecular weight heparin for patients with an INR < 1.5 are allowed
* No concurrent agents with proarrhythmic potential, including any of the following: terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, flecainide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Laurie, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was centrally activated on November 10, 2006 and the study was closed to accrual on September 10, 2010. Patients were recruited from 9 cancer clinics in Canada
Period: Overall Study
Arm/Group | Treatment (Sunitinib Malate)
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 patient was cancelled due to intercurrent illness and another 3 were found to be ineligible after review. Those 4 patients were excluded from all analyses.
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 29
Region of Enrollment [Number; unit: participants]
  Canada | 35

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Partial and Complete) Per RECIST
Description: Number of patients who had objective responses after radiology review
Time Frame: Up to 3 years
Population: 1 cancelled patient and 4 ineligible patients were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 35
participants | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 21/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=35)
Hospitalization for Grade 3 hemorrhage (Blood and lymphatic system disorders) | 1
Hospitalization for Grade 3 bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for Grade 3 dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hospitalization for Grade 3 cough (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for Grade 3 fatigue (General disorders) | 1
Grade 4 pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalized for grade 3 edema (Blood and lymphatic system disorders) | 1
Grade 3 infection with normal ANC (Infections and infestations) | 1
Grade 3 hyperkalemia (Investigations) | 1
Hospitalization for Grade 2 fatigue (General disorders) | 1
Grade 2 Esophagitis (Gastrointestinal disorders) | 1
Grade 2 Hypothyroidism (Endocrine disorders) | 1
Grade 3 thrombosis/thrombus/embolism (Vascular disorders) | 1
Hospitalized for grade 3 diarrhea (Gastrointestinal disorders) | 2
Grade 2 Infection with normal ANC (Infections and infestations) | 1
Grade 2 flatulence (Gastrointestinal disorders) | 1
Hospitalized for grade 2 cough (Respiratory, thoracic and mediastinal disorders) | 1
Grade 2 dizziness (Nervous system disorders) | 1
Grade 4 thrombocytopenia (Vascular disorders) | 1
Grade 2 left ventricular systolic dysfunction (Cardiac disorders) | 1
Grade 2 tinnitus (Ear and labyrinth disorders) | 1
Death not associated with CTCAE term (General disorders) | 2
Hospitalization for grade 3 pain (General disorders) | 1
Hospitalized for grade 2 seizure (Nervous system disorders) | 1
Grade 5 infection with unknown ANC (Infections and infestations) | 1
Hospitalization for Grade 3 dehydration (Gastrointestinal disorders) | 1
Hospitalization for grade 4 malignant pericardial effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hospitalized for grade 3 pulmonary/upper respiratory other - subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for grade 4 obstruction/stenosis of airway - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for pleural effusion grade 3 (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for Grade 4 dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Grade 2 hypertension (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=35)
Rhinitis (Immune system disorders) | 2
Hypertension (Cardiac disorders) | 10
Fatigue (General disorders) | 34
Fever (General disorders) | 4
Insomnia (General disorders) | 11
Rigors/chills (General disorders) | 4
Sweating (General disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6
Hand-foot (Skin and subcutaneous tissue disorders) | 8
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 12
Dermatology - Other (Skin and subcutaneous tissue disorders) | 7
Hypothyroidism (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 23
Constipation (Gastrointestinal disorders) | 18
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 18
Distension (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 10
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 17
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 24
Taste alteration (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 11
GI - Other (Gastrointestinal disorders) | 2
Hemorrhage pulmonary Bronchopulmonary NOS (Blood and lymphatic system disorders) | 4
Hemorrhage pulmonary Nose (Blood and lymphatic system disorders) | 14
Hemorrhage - Other (Blood and lymphatic system disorders) | 2
Infection with normal ANC Bronchus (Infections and infestations) | 2
Infection with normal ANC Lung (Infections and infestations) | 2
Infection with normal ANC Skin (Infections and infestations) | 2
Edema: limb (Blood and lymphatic system disorders) | 9
Edema: trunk/genital (Blood and lymphatic system disorders) | 4
Muscle weakness Extremity-lowe (Musculoskeletal and connective tissue disorders) | 2
Cognitive disturbance (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 10
Involuntary movement (Nervous system disorders) | 3
Mood alteration Anxiety (Nervous system disorders) | 5
Mood alteration Depression (Nervous system disorders) | 2
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 11
Ocular - Other (Eye disorders) | 2
Pain Abdomen NOS (General disorders) | 17
Pain Back (General disorders) | 10
Pain Bone (General disorders) | 2
Pain Chest/thorax NOS (General disorders) | 19
Pain Extremity-limb (General disorders) | 4
Pain Head/headache (General disorders) | 10
Pain Joint (General disorders) | 8
Pain Muscle (General disorders) | 5
Pain Oral cavity (General disorders) | 2
Pain Throat/pharynx/larynx (General disorders) | 4
Pain Tumor pain (General disorders) | 6
Pain - Other (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Flu-like syndrome (General disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less